CLINICAL TRIAL: NCT06536621
Title: Survey About Practice of Neurosonology in Belgium
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, SCOPPETTUOLO Pasquale, Principal Investigator, MD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: Neurosonology_Survey
Record Dates: First submitted 2024-07-27; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Ultrasound; Neurosonology; NeuroPOCUS
Keywords: Stroke; Critical care; Neuromonitoring; Survey; Neurosonology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasounds are widely employed in almost all medical specialties. In Neurology, the applications are numerous nowadays. There is constant interest in the traditional use of US as well as a growing attention towards the newest and most recent applications in clinical/everyday practice. These applications pertain not only to vascular neurology but also to other fields within this specialty, owing to the non-invasive and bedside availability of this tool.

To achieve this, a high level of expertise is required. Paradoxically, certification of skills is neither required nor mandatory for clinical practice. When examining Belgian centers, a wide disparity in training, indications, and ultrasound use in everyday practice becomes apparent. This discrepancy is not unique to Belgium; it has also been demonstrated throughout the rest of Europe. The European Society of Neurosonology and Cerebral Hemodynamic (ESNCH) has already conducted a survey on this subject, and we would like to replicate it at a national level.

The aim of this survey is to describe the use of ultrasound for neurological diseases in Belgian hospitals and practitioners' familiarity with ultrasound modalities across all indications. Understanding the current state of ultrasound practice in Belgium could help promote more homogeneous and high-quality training, increase educational sessions during national meetings, establish a research network, and facilitate the exchange of internal protocols.

Partipants opinions would be greatly appreciated to better understand Belgian expertise in the field and open discussions about the strengths and limitations of the current situation.

After 4 months from the reception of this email, the online questionnaire will no longer be available, and the investigators will proceed with the analysis of the collected data. As indicated, the inclusion of the hospital name is not mandatory. However, hospital category is kindly request to facilitate our analysis.

Analysis and comparison between categories (such as the type of hospital, region, etc.) will be conducted for research purposes.

For any additional inquiries regarding the survey questions, data collection, and conclusions of the inquiry, please feel free to contact investigators via email at surveyneurosonology@gmail.com.

DETAILED DESCRIPTION:
Ultrasounds are widely employed in almost all medical specialties. In Neurology, the applications are numerous nowadays. There is constant interest in the traditional use of US as well as a growing attention towards the newest and most recent applications in clinical/everyday practice. These applications pertain not only to vascular neurology but also to other fields within this specialty, owing to the non-invasive and bedside availability of this tool.

To achieve this, a high level of expertise is required. Paradoxically, certification of skills is neither required nor mandatory for clinical practice. When examining Belgian centers, a wide disparity in training, indications, and ultrasound use in everyday practice becomes apparent. This discrepancy is not unique to Belgium; it has also been demonstrated throughout the rest of Europe. The European Society of Neurosonology and Cerebral Hemodynamic (ESNCH) has already conducted a survey on this subject, and we would like to replicate it at a national level.

The aim of this survey is to describe the use of ultrasound for neurological diseases in Belgian hospitals and practitioners' familiarity with ultrasound modalities across all indications. Understanding the current state of ultrasound practice in Belgium could help promote more homogeneous and high-quality training, increase educational sessions during national meetings, establish a research network, and facilitate the exchange of internal protocols.

Partipants opinions would be greatly appreciated to better understand Belgian expertise in the field and open discussions about the strengths and limitations of the current situation.

After 4 months from the reception of this email, the online questionnaire will no longer be available, and the investigators will proceed with the analysis of the collected data. As indicated, the inclusion of the hospital name is not mandatory. However, hospital category is kindly request to facilitate our analysis.

Analysis and comparison between categories (such as the type of hospital, region, etc.) will be conducted for research purposes.

For any additional inquiries regarding the survey questions, data collection, and conclusions of the inquiry, please feel free to contact investigators via email at surveyneurosonology@gmail.com.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist in Belgian Hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Practionner of US in Neurology clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Ultrasound (US) centers in Belgium | During four month
  Percentage of hospital centers in Belgium performing ultrasound (US). Number of centers responding to the survey, team and equipment of each center.
  Variable are indicated as numbers and percentage.
Type of US perfomed in the center | During four month
  Number, percentage and subtype (ophtalmic artery, PFO) of extra-cranial and intra-cranial exams for each center. The results are indicated as number and percentage.
Education | During four month
  Information about certification and training of neurosonologist as well as teaching units for residency program.

CONTACTS AND LOCATIONS:
Locations (1):
- Pasquale Scoppettuolo, Brussels, Belgium